CLINICAL TRIAL: NCT06963112
Title: Impact of Intraoperative Midazolam on Delirium Outcome of Elderly Patients (I-IMODE): a Multicentre Randomised Controlled Trial
Brief Title: Intraoperative Midazolam on Delirium Outcome of Elderly Patients
Acronym: IMODE
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: Changhai hospital of Navy Medical University (Unknown); China-Japan Union Hospital, Jilin University (Other); The First Affiliated Hospital of Nanchang University (Other); The First Affiliate Hospital of Guangxi Medical College (Unknown); Second Hospital of Jilin University (Other)
Responsible Party: Principal Investigator, Hao Li, Professor, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PLAGH-IMODE
Record Dates: First submitted 2025-04-09; First posted 2025-05-08 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Delirium; Anxiety
Keywords: midazolam; delirium; anxiety
MeSH Terms: conditions — Delirium; Anxiety Disorders | interventions — Midazolam; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Saline group (Placebo Comparator): The control group patients were given 2 mL physiological saline during anesthesia induction.
  Interventions: Drug: Saline
- Midazolam group (Experimental): The intervention group patients were given 2mg midazolam injection (Jiangsu Enhua Pharmaceutical Co., Ltd.) during anesthesia induction
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Midazolam — The intervention group patients were given 2mg midazolam injection (Jiangsu Enhua Pharmaceutical Co., Ltd.) during anesthesia induction
  Arms: Midazolam group
Drug: Saline — The control group patients were given 2 mL physiological saline.
  Arms: Saline group

SUMMARY:
This study was a multicenter, randomized, double-blind, placebo-controlled trial to treat elderly surgical patients with low-dose midazolam or placebo for anesthesia induction. The incidence of postoperative 7-day delirium was assessed and compared between two groups, to provide valuable reference for clinical practitioners in the use of midazolam in elderly surgical patients.

DETAILED DESCRIPTION:
This study is a multicenter, randomized, double-blind, placebo-controlled trial. A total elderly patients who underwent elective non cardiac surgery were included in the plan and randomly divided into an intervention group and a control group. The intervention group patients were given 2mg midazolam injection (Jiangsu Enhua Pharmaceutical Co., Ltd.) during anesthesia induction; The control group patients were given equal volume physiological saline. Follow up assessment of postoperative delirium and anxiety will be conducted 1-7 days after surgery, and cognitive function follow-up will be conducted 1 month after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. 65 ≤ Age ≤ 85 years old;
2. Elective surgery under general anesthesia, with an estimated surgery time of ≥ 2 hours;
3. Non cardiac surgery, non neurosurgical surgery;
4. ASA grades I-III;
5. Agree to participate and sign the informed consent form;

Exclusion Criteria:

1. Preoperative history of comorbidities such as depression and schizophrenia;
2. History of neurological disorders, moderate stroke;
3. Long term use of benzodiazepines before surgery;
4. 18.5≤BMI≤30 kg/m2
5. There is cognitive impairment, which is determined based on Mini Mental State Examination (MMSE) scores below the standard threshold;
6. There are communication barriers, such as severe dementia, language barriers, and severe hearing or visual impairments;
7. There are any contraindications for the use of midazolam (contraindications for patients with severe respiratory dysfunction, patients with severe liver and kidney damage, patients with sleep apnea syndrome, and patients known to be allergic to benzodiazepines);
8. Preoperative severe liver and kidney dysfunction;
9. Patients expected to enter the ICU after surgery;

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 612 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoeprative delirium | Postoperaitve Day 1-7
  Confusion Assessment Method (CAM) to assess the incidence of postoperative delirium, including four features: acute change or fluctuation course of mental status; inattention; altered level of consciousness; disorganized thinking
Incidence of postoperative anxiety | Postoperaitve Day 1-7
  Generalized Anxiety disorder-7 (GAD-7) scale to assess the incidence of postoperative anxiety, with range from 0 to 21 scores, higher scores indicating more anxious.

SECONDARY OUTCOMES:
Onset time of delirium episodes | Postoperative Day 1-7
  Onset time of delirium episodes
Frequency of delirium episodes | Postoperative Day 1-7
  Frequency of delirium episodes
Subtype of delirium episodes | Postoperative Day 1-7
  Subtype of delirium episodes
Anxiety severity | Postoperative Day 1-7
  GAD-7 scale to assess anxiety severity: 0-4 scores indicating no anxiety, 5-9 scores indicating mild anxiety, 10-14 scores indicating moderate anxiety, ≥15 scores indicating severe anxiety.
Resting and movement pain scores | Postoperative Day 1-3
  Resting and movement pain scores using NRS scale, with the range of 0-10, higher scores indicate more pain.
Intraoperative awareness of the occurrence | Surgery End
  Intraoperative awareness of the occurrence
Incidence of postoeprative nausea and vomiting | Postoperative 1-7
  Incidence of postoeprative nausea and vomiting
Incidence of delayed extubation | Surgery End
  Incidence of delayed extubation
Incidence of non delirium complications and all-cause mortality | Postoperative Day 1-30
  Incidence of non delirium complications and all-cause mortality
Length of hospital stay | Postoperative Day 1-30
  Length of hospital stay
1-Year mortlity | Postoperative 1 year
  1-Year mortlity

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes